CLINICAL TRIAL: NCT03129958
Title: Correlation Between Neck Pain and Postural Abnormalities Among Female Office Workers at University of Dammam
Status: Completed | Type: Observational
Sponsor: Doaa AL-Saleh (Other)
Responsible Party: Sponsor-Investigator, Doaa AL-Saleh, DOAA AL-SALEH, Imam Abdulrahman Bin Faisal University
Organization: Imam Abdulrahman Bin Faisal University (Other)
Other Study IDs: Doaa
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: NECK PAIN
Keywords: NECK PAIN, OFFICE WORKERS
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a cross sectional study conducted to find out the Correlation between neck pain and postural abnormalities among female office workers at University of Dammam by objective assessments methods.

Eligible participants will sign the consent form followed by filling up demographic data, visual analog scale & neck disability index.

After that, Forward Head posture and Thoracic Kyphosis posture will take place by valid and reliable methods.

DETAILED DESCRIPTION:
The study population and sampling were calculated by Raosoft sample size calculator using an estimated average of population size 200 and allowing a 5% tolerable error, based on a 95% confidence interval (CI).

About 140 female office workers were targeted from the medical colleges of University of Dammam (UoD); Medicine, Applied Medical Science, Nursing, Dentistry, Clinical Pharmacology and Health Track of preparatory year were recruited into the study (N=140).

The study was approved by the Institutional Review Board (IRB) at the University of Dammam (IRB-PGS-2015-03-194).

Eligible individuals for this study were informed of the risks and benefits and were asked to read and sign a written consent form.

Participants' confidentiality was maintained by using a code (number) instead of the participant's name on the data collection form.

All data collection forms were saved in a file and secured in a locker & the electronic file saved with password. Only the researcher and the supervisor had an access to them.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with/without non-specific neck pain complaint.
* Age from 28 up to 40 years old.
* At least 25 working hours a week ( at least 2 hours on computer - at least 3 other office working).
* More than 5 years of experience as an office worker.

Exclusion Criteria:

* Subjects who had prolonged absence from work anticipated within the past 12 months.
* Complain of: cervical radiculopathy, migraine, vestibular Dysfunction.
* Had spinal fracture or surgery.
* Pregnancy.
* History of cervical trauma.
* Comorbid medical conditions as cancer, type 1 diabetes, heart disease.

Ages: 28 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: participants been recruited from the medical collages at university of Dammam
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-06-01; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
pain | 2 min
  by VAS
Disability | 5 min
  by Neck Disability Index
Forward head posture | 10 min
  by Myrin's Inclometer/ Goniometer
Thoracic kyphosis | 10 min
  by spinal mouse

CONTACTS AND LOCATIONS:
Overall Officials: DOAA A AL-SALEH, bachelor, Principal Investigator — Imam Abdulrahman Bin Faisal University

IPD SHARING:
Plan to Share IPD: No